CLINICAL TRIAL: NCT04454359
Title: Nutritional Supplement to Improve Physical Performance in Geriatric Day Hospital Participants: a Pilot Study
Brief Title: Multi-nutrient Supplement to Improve Physical Performance in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: Réseau québécois de recherche sur le vieillissement (Unknown); MUHC-Montreal General Hospital Foundation (Unknown)
Responsible Party: Principal Investigator, Stéphanie Chevalier, Associate Professor, McGill University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 15-633-MUHC
Record Dates: First submitted 2020-06-25; First posted 2020-07-01 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Old Age
Keywords: nutritional supplement; loss of autonomy; rehabilitation

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, double-blinded pilot trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Isocaloric placebos of same taste and texture as the experimental supplements
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXP (Experimental): EXP group will ingest a supplement consisting of 1) flavored whey protein isolate with added pure leucine (3 g) diluted in water, twice daily, before breakfast and before bedtime; doses are adjusted per body weight as follows: 20 g, 25 g or 30 g per category of <65 kg, 65-75 kg and >75 kg of body weight respectively. 2) fish oil containing vitamin D, provided as 7.5 mL liquid oil providing 1500 IU vitamin D3 + 1125 mg EPA + 750 mg DHA, to be ingested once daily.
  Interventions: Dietary Supplement: Multi-nutrient supplement
- CTR (Placebo Comparator): Control will ingest an isocaloric placebo consisting of 1) 30 g maltodextrin, twice daily, following the same schedule, and 2) 7.5 mL corn oil, once daily.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Multi-nutrient supplement
  Arms: EXP
Dietary Supplement: Placebo
  Arms: CTR

SUMMARY:
Geriatric Day Hospitals (GDH) of the McGill University Health Centre and l'Institut de Gériatrie de Montreal offer comprehensive rehabilitation programs including physiotherapy and medical care, but no dietetic counselling for the attending frail population at high risk of malnutrition. This study aims to implement a multi-nutrient supplement to further improve nutritional status, physical function and capacity. A whey protein, leucine, vitamin D and omega-3 fatty acid supplement ingested during 16 weeks will be tested versus an isocaloric placebo on measures of physical performance and muscle mass and strength, in GDH participants. The specific objective of this pilot-study is to test feasibility and adherence; pilot data could lead to a larger trial.

DETAILED DESCRIPTION:
RATIONALE Given the high prevalence of malnutrition of the GDH participants and its impact on poor physical performance, providing a nutritional supplement to increase protein, leucine, vitamin D and omega-3 FA intake should complement and optimize the rehabilitation interventions in improving muscle mass, strength and physical performance.

OBJECTIVES

Implementing the proposed nutritional supplement in the routine care of GDH participants will:

1. test the feasibility, acceptance and adherence to the supplement and its safety
2. provide pilot data to test the superiority of the supplement versus an isocaloric placebo on measures of muscle mass, strength, and physical performance.

STUDY DESIGN. This is a randomized, placebo-controlled, double-blinded trial of two parallel arms, conducted on two sites. Eligible participants will be randomly assigned to one of two groups: experimental (EXP) or control (CTR) in a 1:1 ratio. Randomization will be achieved by computer-generated permuted block of four.

INTERVENTION The EXP arm will ingest a multi-nutrient supplement consisting of whey protein + leucine and fish oil + vitamin D and CTR arm will ingest an isocaloric plabebo, during 16 weeks (about 8 weeks during rehabilitation and 8 more weeks after). Outcome assessment will be performed at baseline, week 8 and week 16, except for body composition measured by DXA at baseline and week 16.

OUTCOMES Primary: feasibility Secondary: physical performance, muscle strength, appendicular lean mass Other: dietary intake, physical activity, clinical markers

STATISTICAL ANALYSIS This pilot study is designed to generate data on feasibility, acceptance and compliance to the supplement and is not powered for identifying statistical differences in the secondary outcomes. A sample size of n=40 (20/group) is planned to test feasibility. Data will be reported as medians and 95% CI.

ELIGIBILITY:
Inclusion Criteria:

* participants of Geriatric Day Hospital programs
* able to understand study requirements (Mini Mental State Exam, MMSE >22/30)
* able to read and speak English or French

Exclusion Criteria:

* BMI >35 kg/m2
* glomerular filtration rate <30 mL/min/SA),
* liver or heart failure,
* stroke in the last 6 months (unless totally recovered),
* Parkinson's disease or severe neurologic conditions,
* active malignancies,
* acute inflammation (CRP >10 mg/L),
* known diagnostic of hyperparathyroidism,
* recent acute weight loss (>10% in 3 months, unless stabilized),
* allergy to milk and/or fish,
* long-term use of corticosteroids or anti-neoplastic medication

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-08-10 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
Feasibility: recruitment rate | Recruitment over 2 years
  Recruitment rate (measured in %, compared to expected rates)
Feasibility: adherence to intervention | Over 16 weeks
  Adherence to supplements (measured in %, compared to expected rates)
Feasibility: completion | Over 16 weeks
  Completion of study outcome assessments (measured in %, compared to expected rates)

SECONDARY OUTCOMES:
6-minute walking test | Weeks 0, 8 and 16
  6-minute walking test (measured as the distance walked during 6 minutes, along a 30-m corridor, expressed in m)
Chair stand test | Weeks 0, 8 and 16
  30-second chair stand test: measured as the number of stands from a chair without arms, in 30 sec)
Timed-up-and-go test | Weeks 0, 8 and 16
  Timed-up-and-go (time to get up from a chair without armrest, walk 3 m and return to sit down completely on the chair, measured in seconds)
Handgrip strength | Weeks 0, 8 and 16
  Maximal handgrip strength (using hand-held Jamar dynamometer, measured in kg),
Leg strength | Weeks 0, 8 and 16
  Isometric knee extension peak torque (using Biodex, measured in N)
Appendicular lean mass | Weeks 0 and 16
  Sum of soft lean mass from arms and legs (measured by iDXA, in kg)

OTHER OUTCOMES:
Protein intake | Weeks 0, 8 and 16
  Protein intake (g) from foods and supplements, estimated from 3-day food diary (using Food Processor with Canadian Nutrient File)
Step counts | Weeks 0, 8 and 16
  Measured by accelerometry during 4 days (Actigraph)
Serum albumin | Weeks 0, 8 and 16
  Albumin, in g/L (measured by the MUHC biochemical laboratory)
Serum pre-albumin | Weeks 0, 8 and 16
  Pre-albumin, in mg/L (measured by the MUHC biochemical laboratory)
Serum C-reactive Protein | Weeks 0, 8 and 16
  CRP, in mg/L (measured by the MUHC biochemical laboratory)
Serum Vitamin D | Weeks 0, 8 and 16
  Vitamin D status, 25(OH)D, in nmol/L (measured by the MUHC biochemical laboratory)
Plasma glucose | Weeks 0, 8 and 16
  Glucose, in mmol/L (measured with glucose oxidase method)
Serum IGF-1 | Weeks 0, 8 and 16
  IGF-1, in ng/mL (measured by ELISA)
Plasma phospholipid omega-3 fatty acids | Weeks 0, 8 and 16
  EPA and DHA, expressed as a proportion (%) over total; used as an objective measure of adherence to fish oil supplement (measured by gas chromatography-flame ionization)
Energy intake | Weeks 0, 8 and 16
  energy intake (kcal) from average of 3-day food diary (using Food Processor with Canadian Nutrient File)

CONTACTS AND LOCATIONS:
Overall Officials: Stéphanie Chevalier, PhD, Principal Investigator — Research Institute of the McGill University Health Centre

IPD SHARING:
Plan to Share IPD: No
IPD sharing was not planned originally and therefore consent was not obtained for it.

REFERENCES:
- [Derived] Tessier AJ, Levy-Ndejuru J, Moyen A, Lawson M, Lamarche M, Morais JA, Bhullar A, Andriamampionona F, Mazurak VC, Chevalier S. A 16-week randomized controlled trial of a fish oil and whey protein-derived supplement to improve physical performance in older adults losing autonomy-A pilot study. PLoS One. 2021 Aug 23;16(8):e0256386. doi: 10.1371/journal.pone.0256386. eCollection 2021. PMID 34424934